CLINICAL TRIAL: NCT00125099
Title: Safety and Immunogenicity of the HIV-1 DNA Vaccine VRC-HIVDNA009-00-VP (GAG-POL-NEF-MULTICLADE ENV) in HIV-1 Infected Subjects Treated During Acute HIV Infection
Brief Title: Safety of and Immune Response to a DNA HIV Vaccine (VRC-HIVDNA009-00-VP) in HIV Infected Individuals With Acute HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5187; 10010 (Registry Identifier: DAIDS ES Registry Number); ACTG A5187
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Experienced; Treatment Interruption; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: VRC-HIVDNA009-00-VP

SUMMARY:
The purpose of this study is to evaluate whether the HIV vaccine VRC-HIVDNA009-00-VP will be safe in individuals who started antiretroviral therapy during acute HIV-1 infection. The study will also test whether the vaccine can increase the immune system function in these participants.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has greatly improved mortality and morbidity rates associated with HIV and AIDS. However, many HIV-1 infected individuals are unable to access HAART. It is therefore important to develop a safe and effective therapeutic vaccine to improve immune control of viral replication and reduce the need for antiretroviral medication. This study will evaluate the safety and immunogenicity of the HIV-1 DNA vaccine VRC-HIVDNA009-00-VP in treating HIV-1 infected individuals who initiated antiretroviral therapy during acute infection. This study will involve a supervised treatment interruption (STI) in order to determine whether therapeutic vaccination results in improved immune control of viral replication.

Participants in this study will be randomly assigned to receive either the therapeutic vaccine or placebo in addition to their regular HAART regimens. During the first part of the study, participants will receive 4 vaccinations at Weeks 0, 4, 8 and 24. All individuals completing the therapeutic vaccination phase (defined as completing at least 3 immunizations, including the Week 24 immunization) will be given the opportunity to participate in the second part of the study and undergo a supervised discontinuation of HAART. At Week 30, these participants will discontinue all antiretroviral treatment and will be closely monitored. Participants will restart HAART if they experience a significant decline in their CD4 count, an increase in their viral loads, or if their physicians recommend they resume HAART. At Week 52, all other participants can restart HAART at the discretion of their primary physician.

21 study visits will occur over a period of 52 weeks. After Week 52, monthly study visits will occur through Week 72. Study visits will last approximately two hours and will include physical exams and blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Treated acute HIV-1 infection (initiated HAART during the acute retroviral syndrome AND were diagnosed by a positive HIV-1 viral load and a negative or indeterminate Western blot)
* Minimum of 6 months of HAART, defined as 2 or more antiretroviral drugs in combination
* At least three CD4 cell counts over 350 cells/mm3 for a period of 6 months prior to study entry
* Screening CD4 cell count over 350 cells/mm3 within 30 days prior to study entry
* HIV-1 RNA levels over 50 copies/ml for a period of 6 months prior to study entry
* Screening HIV-1 RNA level less than 50 copies/ml within 30 days prior to study entry
* Agrees to use acceptable methods of contraception

Exclusion Criteria:

* History of serious adverse reactions to vaccines
* History of CD4 cell count less than 250 cells/mm3, opportunistic infections, or AIDS-defining illnesses. Patients who have had one CD4 count less than 250 cells/mm3 or who have had CD4 counts less than 250 cells/mm3 for not more than 2 weeks during acute infection are not excluded.
* History of autoimmune disease, immunodeficiency, asthma, diabetes requiring insulin or oral hypoglycemics, thyroid disease, bleeding disorder, active malignancy, viral hepatitis, or asplenia
* Positive HBV, HCV, or syphilis test
* Suspected allergy or adverse reaction to any component of the study agent
* Changes in antiretroviral regimen within 6 months prior to entry due to virologic failure (not including toxicities)
* Previous participation in STIs
* Pregnancy or breast-feeding
* Live attenuated vaccines or investigational research agents within the 30 days prior to study entry
* Blood products within the 120 days prior to study entry
* Immunoglobulin within the 60 days prior to study entry
* Subunit or killed vaccines or allergy treatments with antigen injections within the 14 days prior to study entry
* Prior experimental HIV vaccines
* Certain immunosuppressive medications within the 6 months prior to study entry
* Current TB prophylaxis or therapy
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization. An individual who has either completed therapy OR is clinically stable for at least 14 days prior to study entry is eligible.
* Anti-dsDNA antibody greater than the upper limit of normal

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Grade 3 or 4 sign/symptom, laboratory abnormality, or death that may be related to the vaccine
2 consecutive viral loads of 400 copies/ml or more while receiving HAART
2 consecutive absolute CD4 cell counts of 250 cells/mm3 or more while receiving HAART
2 consecutive CD4 cell counts more than 50% below the baseline CD4 cell count

SECONDARY OUTCOMES:
Tolerability (receipt of the full schedule of 4 vaccines)
viral load setpoint: average of the log10 viral load measures at Weeks 18, 20, and 22 after HAART withdrawl (study Weeks 48, 50, and 52)
Positive vaccine-elicited ELISPOT response as defined by a twofold increase from baseline that is also 100 or more spots/1,000,000 PBMCs
Positive vaccine-elicited intracellular cytokine staining response as defined by a twofold increase from baseline AND 300 or more spots/1,000,000 PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Dan H. Barouch, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center, Division of Viral Pathogenesis; Eric S. Rosenberg, MD, Study Chair — Massachusetts General Hospital, Division of Infectious Diseases
Locations (5):
- United States (5):
  - Ucsd, Avrc Crs, San Diego, California
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Aaron Diamond AIDS Research Ctr. AIEDRP, New York, New York
  - UW Primary Infection Clinic CRS, Seattle, Washington

REFERENCES:
- [Background] Altfeld M, Rosenberg ES, Shankarappa R, Mukherjee JS, Hecht FM, Eldridge RL, Addo MM, Poon SH, Phillips MN, Robbins GK, Sax PE, Boswell S, Kahn JO, Brander C, Goulder PJ, Levy JA, Mullins JI, Walker BD. Cellular immune responses and viral diversity in individuals treated during acute and early HIV-1 infection. J Exp Med. 2001 Jan 15;193(2):169-80. doi: 10.1084/jem.193.2.169. PMID 11148221
- [Background] Rosenberg ES, Altfeld M, Poon SH, Phillips MN, Wilkes BM, Eldridge RL, Robbins GK, D'Aquila RT, Goulder PJ, Walker BD. Immune control of HIV-1 after early treatment of acute infection. Nature. 2000 Sep 28;407(6803):523-6. doi: 10.1038/35035103. PMID 11029005
- [Result] Rosenberg ES, Graham BS, Chan ES, Bosch RJ, Stocker V, Maenza J, Markowitz M, Little S, Sax PE, Collier AC, Nabel G, Saindon S, Flynn T, Kuritzkes D, Barouch DH; AIDS Clinical Trials Group A5187 Team. Safety and immunogenicity of therapeutic DNA vaccination in individuals treated with antiretroviral therapy during acute/early HIV-1 infection. PLoS One. 2010 May 10;5(5):e10555. doi: 10.1371/journal.pone.0010555. PMID 20479938